CLINICAL TRIAL: NCT01795183
Title: The Effectiveness and Safety of Amisulpride in Chinese Patients With Schizophrenia - A Prospective Open-Label Multicenter Study
Brief Title: Effectiveness and Safety of Amisulpride in Chinese Patients With Schizophrenia
Acronym: ESCAPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMISUL06155; U1111-1131-0692 (Other: UTN)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amisulpride (Experimental): Patients are treated with Amisulpride referring to the dosage and usage section in Chinese Solian® PI. Amisulpride dosage is adjusted based on individual response and reaches the sufficiency within 1 week
  Interventions: Drug: AMISULPRIDE

INTERVENTIONS:
Drug: AMISULPRIDE — Pharmaceutical form: tablet Route of administration: oral
  Other Names: Solian

SUMMARY:
Primary Objective:

To evaluate the effectiveness of amisulpride in Chinese patients with schizophrenia

Secondary Objective:

To evaluate the overall safety of amisulpride in Chinese patients with schizophrenia.

DETAILED DESCRIPTION:
The study duration by subject will include a 8-week treatment period with 3 follow-up visits.

ELIGIBILITY:
Inclusion criteria :

* Satisfying International Classification of Disease-10 (ICD) diagnostic criteria of schizophrenia;
* Positive and Negative Syndrome Scale (PANSS) total score ≥ 60

Exclusion criteria:

* Refractory schizophrenia or Patients treated with sufficient clozapine for a minimum period of 6-8 weeks without improvement;
* Participation into another clinical trial within the last month;
* Patients previously or currently treated with amisulpride;
* Patients receiving clozapine within the past 1 month or treated with long-acting formulation of antipsychotic medication within the past 2 months;
* Patients receiving electric convulsive therapy or physical therapy within the past 1 month;
* Patients with coexisting severe systemic diseases;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effective percentage (PANSS score reduced rate≥50%) | Week 8

SECONDARY OUTCOMES:
Early response rate (PANSS score reduced rate: at least 20%) | week 2
Positive and Negative Syndrome Scale (PANSS)-total score improvement | Baseline, Week 8
Clinical Global Impression Scale- Improvement (CGI-I) | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Beijing, China

REFERENCES:
- [Derived] Liang Y, Yu X. Effectiveness of amisulpride in Chinese patients with predominantly negative symptoms of schizophrenia: a subanalysis of the ESCAPE study. Neuropsychiatr Dis Treat. 2017 Jun 28;13:1703-1712. doi: 10.2147/NDT.S140905. eCollection 2017. PMID 28721051
- [Derived] Liang Y, Yu X. The effectiveness and safety of amisulpride in Chinese patients with schizophrenia who switch from risperidone or olanzapine: a subgroup analysis of the ESCAPE study. Neuropsychiatr Dis Treat. 2017 Apr 21;13:1163-1173. doi: 10.2147/NDT.S132363. eCollection 2017. PMID 28461752